CLINICAL TRIAL: NCT01048866
Title: A Repeat-Dose, Multi-Centre, Randomized, Double-Blind, Placebo-Controlled, Study to Determine the Safety and Efficacy of Flurbiprofen 8.75 mg Lozenge Compared to Its Vehicle Control Lozenge in Patients With Painful Pharyngitis
Brief Title: A Study of Flurbiprofen 8.75 mg Lozenge in Patients With Pharyngitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TH 0913
Record Dates: First submitted 2010-01-13; First posted 2010-01-14 (Estimated); Results first posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Pharyngitis
Keywords: pharyngitis; swollen throat; difficulty swallowing
MeSH Terms: conditions — Pharyngitis; Deglutition Disorders | interventions — Flurbiprofen; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- flurbiprofen 8.75 mg lozenge (Experimental): Participants were instructed to suck one study (flurbiprofen 8.75 mg) lozenge and efficacy assessments were taken in the clinic. Upon discharge, participants were instructed to use another study medication lozenge every 3-6 hours, up to a total of 5 study lozenges in 24 hours. Following efficacy assessments, participants were again instructed to use study medication lozenge every 3-6 hours, up to a total of 5 study lozenges per day (plus rescue medication if needed) for the remaining time in the 7 day study.
  Interventions: Drug: flurbiprofen; Drug: acetaminophen 650mg
- placebo lozenge (Placebo Comparator): Participants were instructed to suck one study (placebo) lozenge and efficacy assessments were taken in the clinic. Upon discharge, participants were instructed to use another lozenge every 3-6 hours, up to a total of 5 study lozenges in 24 hours. Following efficacy assessments, participants were again instructed to use a lozenge every 3-6 hours, up to a total of 5 study lozenges per day (plus rescue medication if needed) for the remaining time in the 7 day study.
  Interventions: Drug: placebo; Drug: acetaminophen 650mg

INTERVENTIONS:
Drug: placebo — Sugar-based lozenge flavoured to match the active treatment lozenge. Instructions were to suck one lozenge until gone, every 3-6 hours as needed for sore throat pain. The participant took nothing by mouth except study medication during the first two hours while at the site. For each re-dosing during the remaining time in the study, alcohol and caffeine-containing beverages (e.g., coffee, tea, hot chocolate, caffeinated soft drinks) were not consumed within 1 hour before the participant used a study medication lozenge.
  Arms: placebo lozenge
Drug: flurbiprofen — Sugar-based, flavoured flurbiprofen 8.75 mg lozenge. Instructions were to suck one lozenge until gone, every 3-6 hours as needed for pain. The participant took nothing by mouth except study medication during the first two hours while at the site. For each re-dosing during the remaining time in the study, alcohol and caffeine-containing beverages (e.g., coffee, tea, hot chocolate, caffeinated soft drinks) were not consumed within 1 hour before the participant used a study medication lozenge.
  Arms: flurbiprofen 8.75 mg lozenge
Drug: acetaminophen 650mg — Rescue medication to be taken as needed. Rescue medication was not blinded.
  Other Names: Tylenol

SUMMARY:
The purposes of this study is to demonstrate the analgesic efficacy of flurbiprofen 8.75 mg lozenge compared to its vehicle lozenge and to demonstrate the safety of the flurbiprofen lozenge throughout the course of treating sore throat due to acute pharyngitis.

DETAILED DESCRIPTION:
Per randomization to the treatments and under double-blind conditions, patients were instructed to suck 1 sugar-based, flavoured flurbiprofen 8.75 mg lozenge or 1 sugar-based, flavoured matching vehicle control/placebo lozenge and remained at the study center for a 2-hour observation period to assess their responses to the study medication during the initial 2-hour post-dose period. Patients were allowed a dose of rescue medication (acetaminophen 650mg), as needed, post-treatment dosing during the study.

After the initial 2 hours in the research center, patients were discharged with an outpatient diary to continue (while awake) to document hourly assessments of Sore Throat Pain Intensity Scale (STPIS), Difficulty Swallowing Scale (DSS), and Swollen Throat Scale (SwoTS) through 24 hours. They used the assigned lozenges as needed every 3-6 hours, up to 5 lozenges over 24 hours. A Follow-Up Visit was conducted for the 24-hour assessments.

Patients received additional study lozenges for use as needed (up to 5 lozenges per 24 hours) over the following 6 days, rescue medication (acetaminophen 650 mg) and a Diary to document their safety and efficacy assessments immediately before and postdose after each as-needed use of a lozenge for the remaining days in the 7-day treatment period. At the end of the 7-day trial, patients returned to the research center for final assessments, review of adverse events over the week, and discharge from the study.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a complaint of sore throat.
2. If the patient is a female of childbearing potential, she has been using effective contraception since the last date of menses and is not breast-feeding or lactating.
3. If the patient is a female of childbearing potential, the patient must have a negative urine pregnancy.
4. The patient has provided written informed consent prior to any study-related procedures.

Exclusion Criteria:

1. The patient has a history of an upper gastrointestinal ulcer within the past 60 days, is currently experiencing clinically significant upper gastrointestinal complaints, or is currently taking medication regularly (≥ three times in the previous week).
2. The patient has a history of any hepatic disease or renal dysfunction.
3. The patient has a history of chronic analgesic use (≥ three times per week over the prior four weeks). (Patients on low-dose aspirin therapy may be allowed in the study per investigator's clinical decision.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-11; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J Shea, BS, Study Director — Reckitt Benckiser Inc.
Locations (1):
- Bluestone Center for Clinical Research, New York, New York, United States

REFERENCES:
- [Result] Schachtel B, Aspley S, Berry P, Muir N, Shephard A, Shea T, Smith G, Schachtel E. Efficacy of a novel (lozenge) delivery of flurbiprofen over 24 hours. Journal of Pain 2012;13(4)Supplement:S74.
- [Result] Aspley S, Schachtel B, Berry P, Shephard A, Shea T, Smith G, Lorton M, Schachtel E. Efficacy and safety of multiple uses of flurbiprofen 8.75mg lozenge over 1 week. Abstract presented at the 14th World Congress on Pain, 27 - 31 August 2012, Milan.
- [Result] Shephard A, Smith G, Aspley S, Schachtel B. Efficacy of flurbiprofen 8.75 mg lozenges for streptococcal and non-streptococcal sore throat: pooled analysis of two randomised, placebo-controlled studies. Abstract presented at the European Congress of Clinical Microbiology and Infectious Diseases (ECCMID), 27 - 30 April 2013, Berlin.
- [Result] Shephard A, Smith G, Aspley S, Schachtel B. Symptomatic relief in streptococcal and non-streptococcal sore throat patients: pooled analysis of two randomised, placebo-controlled studies. Abstract presented at the European Congress of Clinical Microbiology and Infectious Diseases (ECCMID), 27-30 April 2013, Berlin.
- [Result] Schachtel B, Aspley S, Berry P, Shephard A, Sanner K, Shea T, Smith G, Schachtel E. Chief Complaint: the therapeutogenic stimulus as the primary, individualized endpoint in clinical trials. Journal of Pain 2012;13(4)Supplement:S6.
- [Derived] Shephard A, Smith G, Aspley S, Schachtel BP. Randomised, double-blind, placebo-controlled studies on flurbiprofen 8.75 mg lozenges in patients with/without group A or C streptococcal throat infection, with an assessment of clinicians' prediction of 'strep throat'. Int J Clin Pract. 2015 Jan;69(1):59-71. doi: 10.1111/ijcp.12536. Epub 2014 Oct 9. PMID 25296661
- [Derived] Schachtel B, Aspley S, Shephard A, Shea T, Smith G, Schachtel E. Utility of the sore throat pain model in a multiple-dose assessment of the acute analgesic flurbiprofen: a randomized controlled study. Trials. 2014 Jul 3;15:263. doi: 10.1186/1745-6215-15-263. PMID 24988909

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three hundred and thirty-six patients were screened.
Groups:
- Flurbiprofen 8.75 mg Lozenge: Participants were instructed to suck one study (flurbiprofen 8.75 mg) lozenge every 3-6 hours, up to a total of 5 study lozenges in 24 hours for the 7 days of the study. Rescue medication (acetaminophen 650mg) was allowed as needed.
- Placebo Lozenge: Participants were instructed to suck one study (placebo) lozenge every 3-6 hours, up to a total of 5 study lozenges in 24 hours for the 7 days of the study. Rescue medication (acetaminophen 650mg) was allowed as needed.
Period: Overall Study
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Started | 101 | 97
Completed | 97 | 92
Not Completed | 4 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 0 | 2
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge | Total
Number analyzed (Participants) | 101 | 97 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.5 (11.03) | 34.2 (11.17) | 33.9 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 119
  Male | 40 | 39 | 79
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 10 | 10 | 20
  Black or African | 13 | 14 | 27
  White | 67 | 67 | 134
  Multi-racial (no primary) | 3 | 3 | 6
  Other, not specified | 8 | 3 | 11
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 16 | 10 | 26
  Non-Hispanic or non-Latino | 85 | 87 | 172
Sore Throat Pain Intensity Scale (STPIS) [Mean (Standard Deviation); unit: units on a scale] — STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain.
  units on a scale | 79.1 (8.09) | 79.1 (8.37) | 79.1 (8.21)
Difficulty Swallowing Scale (DSS) [Mean (Standard Deviation); unit: units on a scale] — DSS measures difficulty swallowing (dysphagia) using a 100-mm visual analog scale completed by participants. Participants were instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated not difficult and 100-mm indicated very difficult.
  units on a scale | 77.9 (10.55) | 78.2 (10.3) | 78.0 (10.45)
Swollen Throat Scale (SwoTS) [Mean (Standard Deviation); unit: units on a scale] — SwoTS measures how swollen a participant's throat felt using a 100-mm visual analog scale completed by participants. Participants were instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen.
  units on a scale | 76.0 (12.90) | 76.0 (12.7) | 76.0 (12.80)

OUTCOME MEASURES:

1. Primary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale (STPIS) Over the 24 Hours Post-baseline (STPIS SPID24)
Description: STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain. SPID24 was calculated as the sum of the time weighted pain intensity differences from baseline until 24 hours. The full range was -104412 (complete pain relief within 1 hour of dosing that lasts 24 hours) to 27588 (maximum pain within 1 hour lasting 24 hours) using the mean baseline STPIS.
  Participants with a last recorded time point <21 hours were considered Not Evaluable. If a participant used rescue medication, all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments were imputed using linear interpolation assuming the time of the missing assessment to be the nominal time since initial dose.
Time Frame: baseline (pre-dose), post-dose - hourly up to 24 hours
Population: Intent to treat population of participants who took the first full dose of medication, and had STPIS values recorded >= 21 hours post initial dose. Four participants (2 Flurbiprofen, 2 placebo) did not have sufficient 24 hour data to be included in the primary analysis of the primary endpoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 99 | 95
units on a scale | -522.9 (476.54) | -326.5 (386.83)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0021, ANOVA — The a priori threshold for statistical significance is 0.05; least-square means difference = -196.6, 95% CI 2-sided [-321.0 to -72.2]

2. Secondary Outcome: Time Weighted Summed Differences in Difficulty Swallowing Scale (DSS) During the Initial 2 Hours From Baseline
Description: DSS measures difficulty swallowing (dysphagia) using a 100-mm visual analog scale completed by participants. Participants were instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated not difficult and 100-mm indicated very difficult.
  Data are reported as the sum of the time-weighted pain intensity differences from baseline until 2 hours post dose. The full range was -9360 (no difficulty swallowing within 1 hour of dosing that lasts 2 hours) to 2640 (maximum difficulty swallowing within 1 hour of dosing lasting 2 hours) using the baseline DSS value.
  Missing values of DSS with non-missing values at assessments before and after were calculated using linear interpolation.
Time Frame: Baseline (pre-dose), Hours 1 and 2 post-dose
Population: Intent to treat population of participants who took the first full dose of medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
units on a scale | -37.1 (39.60) | -18.1 (29.43)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0002, ANOVA — The a priori threshold for statistical significance is 0.05; Baseline DSS fitted as a covariate and centre as a fixed effect; least-square means difference = -19.0, 95% CI 2-sided [-28.7 to -9.3]

3. Secondary Outcome: Time Weighted Summed Differences in Difficulty Swallowing Scale (DSS) During the Initial 24 Hours From Baseline
Description: DSS measures difficulty swallowing (dysphagia) using a 100-mm visual analog scale completed by participants. Participants were instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated not difficult and 100-mm indicated very difficult.
  Data are reported as the sum of the time-weighted pain intensity differences from baseline until 24 hours post dose. The full range was -102960 (no difficulty swallowing within 1 hour of dosing that lasts 24 hours) to 29040 (maximum difficulty swallowing within 1 hour of dosing lasting 24 hours) using the baseline DSS value. Negative values indicate improvement in difficulty swallowing.
  Missing values of DSS with non-missing values at assessments before and after were calculated using linear interpolation.
Time Frame: Baseline (pre-dose), hourly readings to 24 hours post-dose
Population: Intent to treat population. Four participants (2 Flurbiprofen and 2 placebo) did not have DSS recorded after 21 hours and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 99 | 95
units on a scale | -555.5 (494.04) | -379.4 (397.66)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0054, ANOVA — The a priori threshold for statistical significance is 0.05; least-square means difference = -179.7, 95% CI 2-sided [-305.7 to -53.8]

4. Secondary Outcome: Time Weighted Summed Differences in Swollen Throat Scale (SwoTS) During the Initial 2 Hours From Baseline
Description: SwoTS measures how swollen a participant's throat felt using a 100-mm visual analog scale completed by participants. Participants were instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen.
  The full range of the sum of the time-weighted swollen throat differences from baseline until 2 hours was -9120 (throat did not feel swollen at all within 1 hour of dosing and lasted 2 hours) to 2880 (maximum swollen throat reported within 1 hour and lasting 2 hours) using the mean baseline SwoTS.
  Negative values for the differences indicate improvement. Missing values of SwoTS with non-missing values at assessments before and after were calculated using linear interpolation.
Time Frame: Baseline (pre-dose), hourly readings to 2 hours post-dose
Population: Intent to treat population of participants who took the first full dose of medication
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
units on a scale | -35.5 (38.92) | -16.9 (29.10)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0008, ANOVA — The a priori threshold for statistical significance is 0.05; least-square means difference = -16.4, 95% CI 2-sided [-25.9 to -7.0]

5. Secondary Outcome: Time Weighted Summed Differences in Swollen Throat Scale (SwoTS) During the Initial 24 Hours From Baseline
Description: SwoTS measures how swollen a participant's throat felt using a 100-mm visual analog scale completed by participants. Participants were instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen.
  The full range of the sum of the time-weighted swollen throat differences from baseline until 24 hours was -100320 (throat did not feel swollen at all within 1 hour of dosing and lasted 24 hours) to 31680 (maximum swollen throat reported within 1 hour and lasting 24 hours) using the mean baseline SwoTS. Negative values for differences indicate improvement.
Time Frame: Baseline (pre-dose), hourly readings to 24 hours post-dose
Population: Intent to treat population. Four participants (2 Flurbiprofen, 2 Vehicle) did not have SwoTS recorded after 21 hours and were not included in the analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 99 | 95
units on a scale | -542.4 (487.67) | -377.4 (419.95)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0087, ANOVA; least-square means difference = -168.4, 95% CI 2-sided [-293.7 to -43.1]

6. Secondary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale (STPIS) Over the 2 Hours Post-baseline (STPIS SPID2)
Description: STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain. SPID2 was calculated as the sum of the time weighted pain intensity differences from baseline until 2 hours post dose. The full range was -9492 (complete pain relief within one hour of dosing that lasts 2 hours) to 2508 (maximum pain within 1 hour lasting 2 hours) using the mean baseline STPIS.
  If a participant used rescue medication (acetaminophen 650mg was allowed as needed post dose), all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments (recorded or derived due to rescue) were imputed using linear interpolation assuming the time of the missing assessment to be the nominal time since initial dose.
Time Frame: baseline (pre-dose), post-dose: 1 hour, 2 hours
Population: Intent to treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
units on a scale | -37.1 (37.04) | -17.9 (26.54)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p < 0.0001, ANOVA; Baseline STPIS fitted as a covariate and centre as a fixed effect; least-square means difference = -19.0, 95% CI 2-sided [-28.0 to -10.0]

7. Secondary Outcome: Time Weighted Sum of Pain Intensity Differences (SPID) in Sore Throat Pain Intensity Scale Over 24 Hours Post-baseline (STPIS SPID24) For Participants With Baseline Practitioner's Assessment of Pharyngeal Inflammation (PAIN) of Moderate or Severe
Description: STPIS measures sore throat pain intensity on a 100-mm visual analog scale completed by participants. A mark at 0-mm indicates no pain upon swallowing and 100-mm indicates severe pain. For the subgroup of patients with moderate/severe pharyngeal inflammation at baseline, SPID24 was calculated as the sum of the time weighted pain intensity differences from baseline until 24 hours. Taking inclusion criteria into account, the full range was -115695 (no pain at any post-dose time (0) - average baseline) to 28505 (maximum possible pain (100) - average baseline).
  Participants with their last recorded time point <21 hours were considered Not Evaluable. If a participant used rescue medication, all post-rescue STPIS values in the 24-hour interval were assigned the baseline value for STPIS. Missing scores of STPIS with non-missing STPIS scores at earlier and later assessments were imput
Time Frame: baseline (pre-dose), 24 hours post dose (measured each hour post dose)
Population: Intent to treat population of participants who took the first full dose of medication and had moderate or severe pharyngeal inflammation at baseline.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 57 | 57
units on a scale | -476.9 (492.12) | -351.3 (425.98)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.1844, ANOVA; Baseline STPIS fitted as a covariate and centre as a fixed effect; least-square means difference = -118.9, 95% CI 2-sided [-295.3 to 57.5]

8. Secondary Outcome: Sore Throat Relief As Reported by Participants 2 Hours After Initial Dose
Description: Participants graded the relief of his/her sore throat at 2 hours post initial dose using the Sore Throat Relief Rating Scale (STRRS), which is a 6-category relief scale.
  The patient was instructed to swallow and asked:
  "Considering how your throat felt before you took the study medicine, circle the phrase that best describes the relief of your sore throat now." Responses were no relief, slight, mild, moderate, considerable, and complete relief.
Time Frame: 2 hours
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
percentage of participants
  No relief | 9.9 | 38.1
  Slight relief | 28.7 | 22.7
  Mild relief | 27.7 | 17.5
  Moderate relief | 17.8 | 18.6
  Considerable relief | 15.8 | 3.1
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Investigators' Clinical Assessment (CLIN) Of Study Medication as a Treatment for Sore Throat at 24 Hours After Initial Dose
Description: Investigators assessed the effectiveness of study medication on the patient's sore throat at 24 hours following initial dose by answering the following question: "Considering the patient's response to the study medicine over the past 24 hours, how do you rate the study medicine as a treatment for sore throat?" Responses were poor, fair, good, very good or excellent.
Time Frame: 24 hours
Population: Intent to treat population. CLIN was not performed for 3 participants (1 Flurbiprofen, 2 placebo).
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 100 | 95
percentage of participants
  Poor | 25.0 | 25.3
  Fair | 27.0 | 29.5
  Good | 26.0 | 24.2
  Very Good | 14.0 | 12.6
  Excellent | 8.0 | 8.4
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.8827, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Participant Satisfaction Score 24 Hours After Initial Dose
Description: After 24 hours of treatment, participants rated their satisfaction with the treatment on a 7-step scale from extremely dissatisfied to extremely satisfied.
Time Frame: 24 hours
Population: Intent to treat population. One placebo participant did not complete a Patient Satisfaction Score.
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 96
percentage of participants
  Extremely dissatisfied | 4.0 | 5.2
  Very dissatisfied | 4.0 | 9.4
  Dissatisfied | 10.9 | 14.6
  Somewhat satisfied | 27.7 | 32.3
  Satisfied | 23.8 | 26.0
  Very satisified | 24.8 | 7.3
  Extremely satisfied | 5.0 | 5.2
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0105, Wilcoxon (Mann-Whitney); Stratified by centre

11. Secondary Outcome: Investigators' Clinical Assessment (CLIN) Of Study Medication as a Treatment for Sore Throat at End of Study (Day 7)
Description: Investigators assessed the effectiveness of study medication on the patient's sore throat at the end of study by answering the following question: "Considering the patient's response to the study medicine over the past 7 days, how do you rate the study medicine as a treatment for sore throat?" Responses were poor, fair, good, very good or excellent.
Time Frame: Day 7 (end of study)
Population: Intent to treat population of participants who completed the study. CLIN was missing for one flurbiprofen participant.
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 96 | 92
percentage of participants
  Poor | 19.8 | 25.0
  Fair | 22.9 | 26.1
  Good | 24.0 | 20.7
  Very Good | 26.0 | 22.8
  Excellent | 7.3 | 5.4

12. Secondary Outcome: Post 24 Hour, Multiple Dose Results: Weighted Sum of Pain Intensity Differences (SPID) Over 2 Hours for the Sore Throat Pain Intensity Scale (STPIS SPID2)
Description: The time weighted summed differences over 2 hours after taking a lozenge after the initial 24-hours post-baseline.
  STPIS is a validated 100-mm visual analog scale completed by participants that measures "pain on swallowing" (odynophagia). A mark at 0-mm indicates no pain and 100-mm indicates severe pain. SPID2 was calculated as the sum of the time-weighted pain intensity differences from a measurement taken prior to taking a lozenge and at hours 1 + 2 after taking the lozenge during Days 2-7. Data for multiple doses/days were averaged to obtain the values used for calculating SPID2. The full range for SPID2 was -5843 to 6157 with negative values indicating improvement in pain intensity. Assessments were summarized using a repeated measures mixed model, with treatment and center as a fixed effect, time since Baseline as a covariate, and a random effect for participants.
Time Frame: Days 2-7
Population: Intent to treat population of participants who were active in the study on day 2. For doses where rescue medication was taken within the 2 hour assessment, all following differences were imputed as zero.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 97 | 92
units on a scale | -22.7 (2.56) | -16.8 (2.61)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0743, ANOVA; Repeated measures ANOVA model with participant as a random effect; least-square means difference = -5.9, 95% CI 2-sided [-12.4 to 0.6]

13. Secondary Outcome: Post 24 Hour, Multiple Dose Results: Weighted Sum of Differences Over 2 Hours for Difficulty Swallowing Scale (DSS2)
Description: The time weighted summed differences over 2 hours after taking a lozenge for all lozenges taken after the initial 24-hours post-baseline.
  To measure the functional effect on pharyngitis, the participant was asked to evaluate his/her difficulty swallowing (dysphagia) using a 100-mm visual analog scale prior to dosing, and 1 hour and 2 hours post dose. The participant was instructed to swallow and "Place a line on the scale that best characterizes how difficult it is to swallow now." A mark at 0-mm indicated not difficult and 100-mm indicated very difficult. Data for multiple doses/days were averaged to obtain the values used for calculating DSS2. The full range for differences was -5626 to 6374 with negative values indicating improvement in pain intensity.
  Assessments were summarized using a repeated measures mixed model, with treatment and center as a fixed effect, time since Baseline as a covariate, and a random effect for participants.
Time Frame: Days 2-7
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 97 | 92
units on a scale | -21.0 (2.49) | -15.5 (2.53)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0871, ANOVA; Repeated measures ANOVA model with patient as a random effect; least-square means difference = -5.5, 95% CI 2-sided [-11.7 to 0.8]

14. Secondary Outcome: Post 24 Hour, Multiple Dose Results: Weighted Sum of Differences Over 2 Hours for Swollen Throat Scale (SwoTS2)
Description: The time weighted summed differences over 2 hours after taking a lozenge for all lozenges taken after the initial 24-hours post-baseline.
  The participant was asked to evaluate how swollen his/her throat felt using a 100-mm visual analog scale prior to dosing, and 1 hour and 2 hours post dose.
  The patient was instructed to swallow and "Place a line on the scale that best characterizes how swollen your throat feels now." A mark at 0-mm indicated not swollen and 100-mm indicated very swollen. Data for multiple doses/days were averaged to obtain the values used for calculating SWoTS2. The full range for differences was -5396 to 6604 with negative values indicating improvement in pain intensity.
  Assessments were summarized using a repeated measures mixed model, with treatment and center as a fixed effect, time since Baseline as a covariate, and a random effect for participants.
Time Frame: Days 2-7
Population: Intent to treat population of participants who were active in the study on day 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 97 | 92
units on a scale | -19.5 (2.49) | -13.4 (2.52)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0595, ANOVA; Repeated measures ANOVA model with participant as a random effect; least-square means difference = -6.0, 95% CI 2-sided [-12.3 to 0.2]

15. Secondary Outcome: Post 24 Hour, Multiple Dose Results: Sore Throat Relief As Reported by Participants 2 Hours After Dosing
Description: Participants graded the relief of his/her sore throat at 2 hours after taking a lozenge for all lozenges taken after the initial 24-hours post-baseline using the Sore Throat Relief Rating Scale (STRRS), which is a 6-category relief scale.
  The patient was instructed to swallow and:
  "Considering how your throat felt before you took the study medicine, circle the phrase that best describes the relief of your sore throat now." Responses following each lozenge were no relief, slight, mild, moderate, considerable, and complete relief. Results summarize responses 2 hours after taking each lozenge.
Time Frame: Days 2-7
Population: Intent to treat population of participants who were active in the study on day 2
Measure: Number; unit: percentage of doses
Units Other Than Participants: Lozenges (doses)
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 97 | 92
Number analyzed (Lozenges (doses)) | 636 | 701
percentage of doses
  No relief | 9.7 | 23.0
  Slight relief | 21.7 | 24.8
  Mild relief | 25.2 | 19.0
  Moderate relief | 16.5 | 13.7
  Considerable relief | 18.9 | 14.7
  Complete relief | 8.0 | 4.9
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0195, ANOVA; Repeated measures ANOVA model with participant as a random effect; least-square means difference = 0.5, 95% CI 2-sided [0.1 to 0.9]

16. Secondary Outcome: Percentage of Participants Who Took Rescue Pain Medication
Description: Participants were allowed a dose of rescue medication (acetaminophen 650mg), as needed, post-treatment dosing during the study.
Time Frame: Days 1-7
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
percentage of participants
  Yes | 13.9 | 25.8
  No | 86.1 | 74.2
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0322, Regression, Logistic; Effect for centre

17. Secondary Outcome: Time to First Rescue Pain Medication
Description: Participants were allowed a dose of rescue medication (acetaminophen 650mg), as needed, post-treatment during the study. Time from initial dose to first rescue medication is summarized by time categories.
Time Frame: Days 1-7
Population: Intent to treat population
Measure: Number; unit: percentage of participants
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
percentage of participants
  2 - <4 hours | 2.0 | 6.2
  4 - <6 hours | 2.0 | 2.1
  6 - <24 hours | 5.9 | 13.4
  24 - <72 hours | 3.0 | 3.1
  72 - 168 hours | 1.0 | 1.0
  Did not rescue | 86.1 | 74.2
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0276, Log Rank

18. Secondary Outcome: Change From Baseline in Body Temperature at 2 Hours Post Initial Dose
Time Frame: baseline (pre-dose), 2 hours post-dose
Population: Safety population
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 101 | 97
degrees Fahrenheit | -0.2 (0.63) | -0.0 (0.82)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.0288, ANOVA; least-square means difference = -0.2, 95% CI 2-sided [-0.4 to -0.0]

19. Secondary Outcome: Change From Baseline in Body Temperature at End of Study
Time Frame: baseline (pre-dose), up to Day 7
Population: Safety population of participants with a recording at the end of study visit.
Measure: Mean (Standard Deviation); unit: degrees Fahrenheit
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Number analyzed (Participants) | 96 | 91
degrees Fahrenheit | -0.4 (0.91) | -0.3 (0.94)
Statistical Analysis 1: Comparison: Flurbiprofen 8.75 mg Lozenge vs Placebo Lozenge; Test type: Superiority or Other; p = 0.4274, ANOVA; least-square means difference = -0.1, 95% CI 2-sided [-0.3 to 0.1]

ADVERSE EVENTS:
Time Frame: Initial dose on Day 1 up to Day 7
Arm/Group | Flurbiprofen 8.75 mg Lozenge | Placebo Lozenge
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/97
Other Adverse Events (participants affected / at risk) | 34/101 | 28/97
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flurbiprofen 8.75 mg Lozenge (N=101) | Placebo Lozenge (N=97)
Lacrimation increased (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0
Gingival erythema (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Oral mucosal erythema (Gastrointestinal disorders) | 0 | 1
Oropharyngeal blistering (Gastrointestinal disorders) | 1 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1
Chills (General disorders) | 1 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Beta haemolytic streptococcal infection (Infections and infestations) | 0 | 1
Conjunctivitis viral (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Otitis externa (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 1 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 1
Headache (Nervous system disorders) | 8 | 6
Migraine (Nervous system disorders) | 0 | 2
Paraesthesia (Nervous system disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal hypoaesthesia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less